CLINICAL TRIAL: NCT03687073
Title: Trial of Indole-3-Carbinol & Silibinin
Brief Title: Trial of Indole-3-Carbinol and Silibinin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS075
Record Dates: First submitted 2018-09-14; First posted 2018-09-27 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — indole-3-carbinol; Silybin; gp100 Melanoma Antigen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single-dose PK study (Experimental): Subjects will take the assigned dose of I3C, Sil, or I3C + Sil once at the study center. Ten mL of blood will be collected at the time points described in Section 9.14. Concurrently, urine will also be collected for 24 hours after the first dose of I3C, Sil or I3C + Sil, divided into the time intervals.
  Interventions: Drug: Indole-3-Carbinol; Drug: Silibinin; Drug: Silibin
- Multi-dose PK Study (Experimental): Subjects will take the assigned dose of I3C, Sil, or I3C + Sil for 8 weeks. Ten mL of blood will be collected at the time points described in Section 9.14. Concurrently, urine will be collected for 24 hours after the first dose of I3C, Sil or I3C + Sil, divided into the time intervals.
  Interventions: Drug: Indole-3-Carbinol; Drug: Silibinin; Drug: Silibin
- Safety Study (Experimental): Safety data will be generated during the multi-dose PK and PD study, as DLT is not anticipated in the single-dose PK study. Enrollment into dose cohorts 1 and 2 can occur on a continuous basis. Enrollment for dose cohorts 3 and 4 will be done sequentially using a modified 3+3 design (see Section 8.2). The first three subjects enrolled into a dose cohort must complete at least 21 days of the multi-dose PK/PD study without a DLT before the remaining 4 subjects in the cohort can be enrolled.
  Interventions: Drug: Indole-3-Carbinol; Drug: Silibinin; Drug: Silibin
- Cohort 4 PD Study (Experimental): The effect of I3C, Sil, or I3C + Sil on the pharmacodynamic endpoints listed under the Secondary Objectives in Section 1.2 will be characterized. This PD study will be done concurrently with the multi-dose PK study. Subjects will take the assigned dose of I3C, Sil, or I3C + Sil for 8 weeks. Nasal epithelium, oral cavity cells, buccal cells, blood, and urine will be collected at the time points described in the study calendar in Section 4.0.
  Interventions: Drug: Indole-3-Carbinol; Drug: Silibinin; Drug: Silibin

INTERVENTIONS:
Drug: Indole-3-Carbinol — Cohorts 2, 3, & 4: 400 mg PO BID
  Other Names: 13C
Drug: Silibinin — Cohorts 1 & 4: 720mg
  Other Names: Sil
Drug: Silibin — Cohort 3: 360mg
  Other Names: Sil

SUMMARY:
This is a non-therapeutic, Phase 1 clinical trial to examine the safety, pharmacokinetic (PK) characteristics, and pharmacodynamics (PD) effect of indole-3-carbinol (I3C) and silibinin (Sil) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Current smoker of ≥ 8 cigarettes per day for at least the last 6 months by self-report
* Adequate blood counts, and adequate liver and kidney function defined as follows:

  * Hemoglobin ≥ 9 g/dL for women, ≥ 10 g/dL for men
  * Platelet count ≥ 100 x 10^9/L
  * Total bilirubin ≤ Institutional upper limit of normal (≤ 1.3 mg/dL for UMMC)
  * ALT ≤ 1.5 times institutional upper limit of normal
  * Creatinine ≤ 1.4 g/dL and estimated GFR ≥ 80 mL/min/1.7m2
* Able to understand the experimental nature of the study and provide informed written consent

Exclusion Criteria:

* Chronic proton pump inhibitor, H2-blocker (i.e., ranitidine, famotidine), and/or calcium carbonate use
* History of gastric bypass surgery, gastric banding, bowel resection, malabsorption syndromes such as celiac sprue or pancreatic insufficiency, or other conditions that may affect gastric or intestinal absorption of nutrients
* Current use of tobacco products other than cigarettes (i.e. snuff, snuz, smokeless tobacco, cigars, pipes), or use of these products within 3 months of study registration
* Major or chronic medical disease, including heart disease, poorly controlled diabetes, etc., to be adjudicated by the principal investigator
* Known active malignancy
* History of aerodigestive malignancies
* Women who are pregnant, intend to become pregnant within 3 months of study registration, or who are lactating. Women of childbearing potential must have a negative urine pregnancy test within 14 days of starting the assigned intervention
* Antibiotic use within 2 months of study registration by self-report
* History of respiratory tract cancer
* Known allergy to I3C, Sil, or its components
* Psychiatric and/or social situations that would potentially limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Safety of the combination of I3C + Sil | Week 8
  Incidence of Dose Limiting Toxicities (DLTs)
Pharmacokinetic profile of I3C + Sil | Week 8
  AUC
Pharmacokinetic profile of I3C + Sil | Week 8
  Cmax
Pharmacokinetic profile of I3C + Sil | Week 8
  Half-life
Pharmacokinetic profile of I3C + Sil | Week 8
  Elimination rate
Pharmacokinetic profile of I3C + Sil | Week 8
  Plasma clearance
Pharmacokinetic profile of I3C + Sil | Week 8
  Renal clearance
Pharmacokinetic profile of I3C + Sil | Week 8
  Accumulation

SECONDARY OUTCOMES:
Effect of I3C, Sil, or I3C + Sil on circulating inflammatory markers | Week 8
  Change in inflammatory markers IL-1B, TNF-a, IL-6, IL-8, Cox-2, prostaglandin E, and C-reactive protein
Effect of I3C, Sil, or I3C + Sil on circulating immunophenotype | Week 8
  Change in circulating immunophenotype
Effect of I3C, Sil, or I3C + Sil on protein expression of phosphorylated-Akt (pAkt), pERK, pSTAT3 and NF-kB from peripheral blood mononuclear cells (PBMC) | Week 8
  Change in protein expression of phosphorylated-Akt (pAkt), pERK, pSTAT3 and NF-kB from peripheral blood mononuclear cells (PBMC)
Effect of I3C, Sil, or I3C + Sil on RNA sequencing from PBMC | Week 8
  Change in of I3C, Sil, or I3C + Sil on
Effect of I3C, Sil, or I3C + Sil on PIK3CA pathway signaling in buccal cells | Week 8
  Change in PIK3CA pathway signaling in buccal cells
Effect of I3C, Sil, or I3C + Sil on PIK3CA pathway signaling in oral cavity cells | Week 8
  Change in PIK3CA pathway signaling in oral cavity cells
Effect of I3C, Sil, or I3C + Sil on PIK3CA pathway signaling in nasal mucosa | Week 8
  Change in PIK3CA pathway signaling in nasal mucosa
Effect of I3C, Sil, or I3C + Sil on fasting glucose | Week 8
  Change in fasting glucose
Effect of I3C, Sil, or I3C + Sil on fasting insulin | Week 8
  Change in fasting insulin
Effect of I3C, Sil, or I3C + Sil on lipid profile | Week 8
  Change in lipid profile
Effect of I3C, Sil, or I3C + Sil on leptin | Week 8
  Change in leptin
Effect of I3C, Sil, or I3C + Sil on body weight | Week 8
  Change in body weight
Effect of I3C, Sil, or I3C + Sil on waist circumference | Week 8
  Change in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fujioka, MD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States